CLINICAL TRIAL: NCT04036968
Title: Evaluating Cannabidiol (CBD) to Enhance the Analgesic Effect of Hydromorphone in Humans
Brief Title: Enhancing Medication-based Analgesia in Humans- STUDY 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB00214289; R01DA040644 (NIH)
Record Dates: First submitted 2019-07-25; First posted 2019-07-30 (Actual); Results first posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Pain; Cannabis; Opioid Use
Keywords: Clinical Trial; Analgesia; Phase II; Abuse potential
MeSH Terms: conditions — Pain; Marijuana Abuse; Agnosia

STUDY DESIGN:
Intervention Model Description: Within-subject study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Study drug administration will be concealed from all study staff and participants to prevent bias in outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo+Placebo (Placebo Comparator): Within-subject double-blind, double-dummy administration of placebo + placebo. Order of dose randomized session days 2-5.
  Interventions: Drug: Within-subject test of blinded study medications
- Hydromorphone+Placebo (Active Comparator): Within-subject double-blind, double-dummy administration of hydromorphone (oral) 4mg + placebo. Always administered during session 1.
  Interventions: Drug: Within-subject test of blinded study medications
- Hydromorphone (oral) 4mg + Cannabidiol 50mg (Experimental): Within-subject double-blind, double-dummy administration of hydromorphone (oral) 4mg + cannabidiol (oral) 50mg. Order of dose randomized session days 2-5.
  Interventions: Drug: Within-subject test of blinded study medications
- Hydromorphone (oral) 4mg + Cannabidiol 100mg (Experimental): Within-subject double-blind, double-dummy administration of hydromorphone (oral) 4mg + cannabidiol (oral) 100mg. Order of dose randomized session days 2-5.
  Interventions: Drug: Within-subject test of blinded study medications
- Hydromorphone (oral) 4mg + Cannabidiol 200mg (Experimental): Within-subject double-blind, double-dummy administration of hydromorphone (oral) 4mg + cannabidiol (oral) 200mg. Order of dose randomized session days 2-5.
  Interventions: Drug: Within-subject test of blinded study medications

INTERVENTIONS:
Drug: Within-subject test of blinded study medications — Within-subject double-blind, double-dummy, study design wherein all participants received all doses in 8-hour outpatient sessions. Primary outcomes assessed during 8-hour outpatient sessions and included laboratory pain testing, subjective reports of drug effects, and cognitive performance, evaluated as a function of study medication condition.

SUMMARY:
This is a single-group, within-subject, double-blind, double-dummy, placebo and active-controlled study evaluated whether the FDA-approved cannabinoid cannabidiol (CBD; Epidiolex) would enhance analgesia, subjective reports, and cognitive performance when compared to the FDA-approved opioid hydromorphone (Dilaudid). This is study 2 is a series of studies.

DETAILED DESCRIPTION:
This was a human laboratory systematic examination of whether adding the FDA-approved cannabinoid cannabidiol (CBD; Epidiolex; oral) to the FDA-approved opioid hydromorphone (Dilaudid; oral) would change the experience of hydromorphone as rated by laboratory measures of pain, subjective reports of drug effects, and cognitive performance. Subjects are healthy individuals with no history of drug use disorder. Study subjects and staff were completed blinded to the study drugs and the class of drugs under investigation and were informed that subjects may receive opioids, stimulants, cannabinoids, benzodiazepines, over the counter medications, and/or placebo. All participants completed all sessions. Sessions lasted up to 8-hours and were conducted at least 7 days apart on an outpatient basis. Primary outcomes were collected from participants prior to dosing and at several hour periods post-dosing.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75
* Urine sample tests negative for common illicit substances of abuse, including cannabis
* Medically cleared to take study medications
* Are not pregnant or breast feeding
* Willing to comply with the study protocol.

Exclusion Criteria:

* Meet DSM-5 criteria for alcohol/substance use disorder
* Taking opioids for pain
* Previous adverse reaction to a cannabinoid product
* Prescribed and taking stimulants or benzodiazepines
* Answer "yes" to item 1 of the Brief Pain Inventory indicating chronic pain
* Self-report any illicit drug or cannabinoid use in the past 7 days
* Presence of any clinically significant medical/psychiatric illness judged by the investigators to put subject at elevated risk for experiencing an adverse event
* History of seizure disorder
* Have a known allergy to the study medications or sesame seed oil
* ALT or AST levels >3x ULN and/or Bilirubin levels >2x ULN during Screening
* Current (past 60-day) suicidal thoughts or past year history of suicidal behavior
* Taking medications contraindicated with hydromorphone or cannabidiol
* Have a history of clinically significant cardiac arrhythmias or vasopastic disease
* Have an abnormal and clinically-significant ECG

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly E Dunn, PhD, Principal Investigator — Johns Hopkins University; Claudia Campbell, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University Bayview Medical Campus, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bergeria CL, Mun CJ, Speed TJ, Huhn AS, Wolinsky D, Vandrey R, Campbell CM, Dunn KE. A within-subject, double-blind, placebo-controlled randomized evaluation of the combined effects of cannabidiol and hydromorphone in a human laboratory pain model. Pain. 2025 Feb 28;166(9):e175-e184. doi: 10.1097/j.pain.0000000000003561. PMID 40839659

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a within-subject study, and all participants (n=31) completed all study conditions. The same 31 participants moved from one treatment arm to the next.
Groups:
- Full Participant Sample: Each participant completed the following five study conditions (arms) in randomized order:
  Placebo + Placebo condition
  Hydromorphone (oral) 4mg + placebo condition
  Hydromorphone (oral) 4mg + Cannabidiol (oral) 50mg condition
  Hydromorphone (oral) 4mg + Cannabidiol (oral) 100mg condition
  Hydromorphone (oral) 4mg + Cannabidiol (oral) 200mg condition
Period: Overall Study
Arm/Group | Full Participant Sample
Started | 31
Placebo + Placebo | 31
Hydromorphoe 4mg + Placebo | 31
Hydromorphone 4mg + Cannabidiol 50mg | 31
Hydromorphone 4mg + Cannabidiol 100mg | 31
Hydromorphone 4mg + Cannabidiol 200mg | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: This is a within group study and same participants went through all treatment arms.
Arm/Group | All Participants
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.3 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 16
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Peak Cold Pressor Tolerance
Description: Peak amount of time participant submerged hand in cold pressor (5 degree circulating cold water) laboratory test of pain as a function of double- blinded study medications (range 0 -300).
Time Frame: 8 hour study session
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Placebo+Placebo | Hydromorphone+Placebo | Hydromorphone (Oral) 4mg + Cannabidiol 50mg | Hydromorphone (Oral) 4mg + Cannabidiol 100mg | Hydromorphone (Oral) 4mg + Cannabidiol 200mg
Number analyzed (Participants) | 31 | 31 | 31 | 31 | 31
minutes | 118.6 (8.8) | 130.8 (8.9) | 161.1 (10.1) | 163.2 (9.9) | 154.6 (9.6)
Statistical Analysis 1: Comparison: Placebo+Placebo vs Hydromorphone+Placebo vs Hydromorphone (Oral) 4mg + Cannabidiol 50mg vs Hydromorphone (Oral) 4mg + Cannabidiol 100mg vs Hydromorphone (Oral) 4mg + Cannabidiol 200mg; Test type: Superiority — Comparison of three drug conditions with cannabidiol to control groups placebo+placebo and hydromorphone+placebo; p = 0.195, ANOVA

2. Primary Outcome: Peak Self-report Rating of "Drug Effect" (0-100), as Measured by the Visual Analog Rating Scale
Description: Peak self-report rating of "Drug Effect" on a 0 ("none at all") to 100 ("extremely") visual analog scale as a function of double- blinded study medication, wherein higher values indicate stronger subjectively-experienced drug effects.
Time Frame: 8 hour study session
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo+Placebo | Hydromorphone+Placebo | Hydromorphone (Oral) 4mg + Cannabidiol 50mg | Hydromorphone (Oral) 4mg + Cannabidiol 100mg | Hydromorphone (Oral) 4mg + Cannabidiol 200mg
Number analyzed (Participants) | 31 | 31 | 31 | 31 | 31
units on a scale | 4.8 (0.7) | 12.6 (1.4) | 15.7 (1.7) | 18.0 (1.6) | 17.9 (1.6)
Statistical Analysis 1: Comparison: Placebo+Placebo vs Hydromorphone+Placebo vs Hydromorphone (Oral) 4mg + Cannabidiol 50mg vs Hydromorphone (Oral) 4mg + Cannabidiol 100mg vs Hydromorphone (Oral) 4mg + Cannabidiol 200mg; Test type: Superiority; p < .001, ANOVA

3. Primary Outcome: Peak Number Accurate on Circular Lights
Description: Peak number accuracy on the Circular Lights fine motor task as a function of double-blinded study drug administration. Participants were provided 60 seconds to press buttons that are lit in randomized order and displayed automatically on a circular lights wall mounted unit. The primary outcome is the number of lit buttons that were accurately pressed within 60 seconds, which is a metric to assess fine motor impairment. Lower numbers are indicative of greater drug-related impairment. There is no upper limit on the circular lights task.
Time Frame: 8 hour study session
Measure: Mean (Standard Error); unit: correct responses
Arm/Group | Placebo+Placebo | Hydromorphone+Placebo | Hydromorphone (Oral) 4mg + Cannabidiol 50mg | Hydromorphone (Oral) 4mg + Cannabidiol 100mg | Hydromorphone (Oral) 4mg + Cannabidiol 200mg
Number analyzed (Participants) | 31 | 31 | 31 | 31 | 31
correct responses | 64.9 (1.0) | 59.2 (1.0) | 64.1 (1.0) | 63.6 (0.9) | 64.3 (0.9)
Statistical Analysis 1: Comparison: Placebo+Placebo vs Hydromorphone+Placebo vs Hydromorphone (Oral) 4mg + Cannabidiol 50mg vs Hydromorphone (Oral) 4mg + Cannabidiol 100mg vs Hydromorphone (Oral) 4mg + Cannabidiol 200mg; Test type: Superiority; p = 0.074, ANOVA

ADVERSE EVENTS:
Time Frame: Up to 40 hours
Description: Adverse events were prompted systematically each hour throughout the session and documented according to good clinical practices. Spontaneously reported adverse events were also documented. All reports of symptoms were categorized as discrete events, such that one experience that included more than 1 symptom would be represented by more than 1 event. Events reported here were all rated as definitely or possibly related to study medication, collapsed across severity (mild, moderate, or severe).
Arm/Group | Placebo+Placebo | Hydromorphone+Placebo | Hydromorphone (Oral) 4mg + Cannabidiol 50mg | Hydromorphone (Oral) 4mg + Cannabidiol 100mg | Hydromorphone (Oral) 4mg + Cannabidiol 200mg
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31 | 0/31 | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 0/31 | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 8/31 | 20/31 | 15/31 | 22/31 | 20/31
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo+Placebo (N=31) | Hydromorphone+Placebo (N=31) | Hydromorphone (Oral) 4mg + Cannabidiol 50mg (N=31) | Hydromorphone (Oral) 4mg + Cannabidiol 100mg (N=31) | Hydromorphone (Oral) 4mg + Cannabidiol 200mg (N=31)
Chills (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Cramp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appetite Decrease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appetite Increase (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Dry Mouth (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 6 (6)
Nausea (Gastrointestinal disorders) | 2 (2) | 6 (6) | 2 (2) | 6 (6) | 7 (7)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Clumsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 5 (5) | 4 (4) | 1 (1)
Drowsiness (Nervous system disorders) | 7 (7) | 13 (13) | 10 (10) | 15 (15) | 15 (15)
Euphoria (Nervous system disorders) | 0 (0) | 5 (5) | 1 (1) | 3 (3) | 1 (1)
Fatigue (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impaired (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Irritability (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Light Headed (Nervous system disorders) | 0 (0) | 3 (3) | 3 (3) | 4 (4) | 5 (5)
Nervousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tingling (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restlessness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shaky (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Yawning (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photosensitivity (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Piloerection (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruitus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dry Eyes (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Frequent Urination (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-18): https://cdn.clinicaltrials.gov/large-docs/68/NCT04036968/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT04036968/ICF_001.pdf